CLINICAL TRIAL: NCT03159455
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 1467335 in Healthy Japanese Male Volunteers With Multiple Oral Doses at the Highest Dose in Caucasian for Comparison (Randomised, Double-blind, Placebo-controlled Trial)
Brief Title: This Study Tests BI 1467335 in Healthy Japanese and Caucasian Men. The Study Tests How Different Doses of BI 1467335 Are Taken up in the Body and How Well They Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1386-0007
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1467335 (Experimental)
  Interventions: Drug: BI 1467335
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1467335 — Duration - 28 days
  Arms: BI 1467335
Drug: Placebo — Duration - 28 days
  Arms: Placebo

SUMMARY:
The primary objective of the current study is to investigate the safety and tolerability of BI 1467335 in healthy Japanese male subjects following oral administration of multiple rising doses The Caucasian group will receive higher dose only.

A secondary objective is the exploration of the pharmacokinetics and pharmacodynamics of BI 1467335 in healthy Japanese and Caucasian male subjects.

ELIGIBILITY:
Inclusion criteria

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP),Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Japanese ethnicity or Caucasian, according to the following criteria:

  * Japanese; born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan
  * Caucasian
* Age of 20 to 45 years (incl.)
* Body Mass Index (BMI) of 18.5 to 25 kg/m2 (incl.) for Japanese and 18.5 to 29.9 kg/m2 (incl.) for Caucasian
* Signed and dated written informed consent by date of Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation.
* Male subjects who agree to minimize the risk of female partners becoming pregnant by fulfilling any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom: combined oral contraceptives, intrauterine device
  * Vasectomised (vasectomy at least 1 year prior to enrolment)
  * Surgically sterilised (including hysterectomy) female partner

Exclusion criteria

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including HIV, viral hepatitis and (or) tuberculosis or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold (or TSPOT) test. Subjects with a positive QuantiFERON TB-Gold (or T-SPOT) test will not participate in the study.
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of biologic agents other than current study medication or drugs considered likely to interfere with the safe conduct of the study
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 half-lives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial (including bioequivalence trial) with an investigational drug within 90 days or 5 half-lives (whichever is greater) prior to planned administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 200 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Have received any live bacterial or live viral vaccination in the 12 weeks prior to the date of screening. Subjects must agree not to receive a live bacterial or live viral vaccination during the study and up to 12 months after the last administration of study drug
* Have received Bacille Calmette-Guerin (BCG) vaccination in the 12 months prior to the date of screening. Subjects must agree not to receive BCG vaccination during the study and up to 12 months after the last administration of study drug
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Signs of cataract at screening by slit lamp test

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-12-16 (Actual); Study Completion 2017-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Souseikai Hakata Clinic, Fukuoka, Fukuoka
  - SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was randomised, double-blind, and placebo-controlled within dose groups. There were 3 sequential dose groups and the highest dose group consisted of 2 ethnic subgroups (Japanese and Caucasian ethnicity).
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated.
Groups:
- Placebo (Japanese): Subjects were orally administered matching placebo tablets with 240 milliliter (mL) water after an overnight fast of at least 10 hours (h) in Japanese ethnicity.
- BI 1467335 3 mg Tablet (Japanese): Subjects were orally administered BI 1467335 3 milligram (mg) film-coated tablets once daily with 240 mL water after an overnight fast of at least 10 h for 28 days in Japanese ethnicity.
- BI 1467335 6 mg Tablet (Japanese): Subjects were orally administered BI 1467335 6 mg film-coated tablets once daily with 240 mL water after an overnight fast of at least 10 h for 28 days in Japanese ethnicity.
- BI 1467335 10 mg Tablet (Japanese): Subjects were orally administered BI 1467335 10 mg film-coated tablets once daily with 240 mL water after an overnight fast of at least 10 h for 28 days in Japanese ethnicity.
- Placebo (Caucasian): Subjects were orally administered matching placebo tablets with 240 mL water after an overnight fast of at least 10 h in Caucasian ethnicity.
- BI 1467335 10 mg Tablet (Caucasian): Subjects were orally administered BI 1467335 10 mg film-coated tablets once daily with 240 mL water after an overnight fast of at least 10 h for 28 days in Caucasian ethnicity.
Period: Overall Study
Arm/Group | Placebo (Japanese) | BI 1467335 3 mg Tablet (Japanese) | BI 1467335 6 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Japanese) | Placebo (Caucasian) | BI 1467335 10 mg Tablet (Caucasian)
Started | 9 | 9 | 9 | 9 | 3 | 9
Completed | 9 | 9 | 9 | 9 | 3 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All subjects who received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Japanese) | BI 1467335 3 mg Tablet (Japanese) | BI 1467335 6 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Japanese) | Placebo (Caucasian) | BI 1467335 10 mg Tablet (Caucasian) | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 3 | 9 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.2 (5.78) | 32.8 (7.16) | 25.0 (6.58) | 25.3 (2.92) | 31.3 (5.86) | 33.7 (5.92) | 29.5 (6.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 9 | 9 | 9 | 9 | 3 | 9 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 9 | 9 | 9 | 3 | 7 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 9 | 9 | 9 | 0 | 0 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 3 | 9 | 12
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events
Description: Percentage of subjects with investigator-defined drug-related Adverse Events (AEs) is reported.
Time Frame: From first day of trial medication intake until end of trial, up to 48 days.
Population: Treated Set (TS): All subjects who received at least 1 dose of trial medication.
Measure: Number; unit: Percentage of subjects
Arm/Group | Placebo (Japanese) | BI 1467335 3 mg Tablet (Japanese) | BI 1467335 6 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Japanese) | Placebo (Caucasian) | BI 1467335 10 mg Tablet (Caucasian)
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 3 | 9
Percentage of subjects | 22.2 | 33.3 | 0.0 | 0.0 | 0.0 | 11.1

2. Secondary Outcome: AUC0-24
Description: Area under the concentration-time curve of BI 1467335 in plasma over the time interval from 0 to 24 hours after administration of the first dose (AUC0-24).
Time Frame: At -0:05 hours (h):minutes (min) before dosing and at 0:15, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00 and 23:55 h:min after first dose.
Population: Pharmacokinetic Set (PKS): This subject set included all subjects of the TS who provide at least 1 pharmacokinetic (PK) parameter that was not excluded due to relevant protocol violations or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/Liter (nmol*h/L)
Arm/Group | BI 1467335 3 mg Tablet (Japanese) | BI 1467335 6 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Caucasian)
Number analyzed (Participants) | 9 | 9 | 8 | 7
nanomole*hour/Liter (nmol*h/L) | 0.898 (69.4) | 2.05 (31.4) | 14.7 (66.9) | 6.39 (33.6)
Statistical Analysis 1: Comparison: BI 1467335 3 mg Tablet (Japanese) vs BI 1467335 6 mg Tablet (Japanese) vs BI 1467335 10 mg Tablet (Japanese); This was non confirmatory testing (Single dose). Dose proportionality of tablets for AUC0-24 was analysed in Japanese subjects; Test type: Other; Slope = 2.2305, 95% CI 2-sided [1.6955 to 2.7655], Standard Error of Mean 0.2592 — Dose proportionality was explored using the power model.The perfect dose proportionality would correspond to a slope β of 1. PK endpoints on the log-transformed scale; Standard error of mean is standard error of slope

3. Secondary Outcome: Cmax
Description: Maximum measured concentration of BI 1467335 in plasma after administration of the first dose (Cmax).
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 3 mg Tablet (Japanese) | BI 1467335 6 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Caucasian)
Number analyzed (Participants) | 9 | 9 | 9 | 9
nanomole/Liter (nmol/L) | 0.791 (60.3) | 1.71 (53.9) | 8.27 (64.5) | 3.42 (55.8)
Statistical Analysis 1: Comparison: BI 1467335 3 mg Tablet (Japanese) vs BI 1467335 6 mg Tablet (Japanese) vs BI 1467335 10 mg Tablet (Japanese); This was non confirmatory testing (Single dose). Dose proportionality of tablets for Cmax was analysed in Japanese subjects; Test type: Other; Slope = 1.9007, 95% CI 2-sided [1.4102 to 2.3912], Standard Error of Mean 0.2382 — [estimate comment as in outcome 2, analysis 1]; Standard error of mean is standard error of slope

4. Secondary Outcome: AUC0-24,28
Description: Area under the concentration-time curve of BI 1467335 in plasma over the time interval from 0 to 24 hours after administration of 28th dose (AUC0-24,28).
Time Frame: At 647:55 hours (h):minutes (min) prior to dosing and at 648:15, 648:30, 648:45, 649:00, 649:30, 650:00, 651:00, 652:00, 654:00, 656:00, 658:00, 660:00 and 672:00 h:min after first drug administration.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/Liter (nmol*h/L)
Arm/Group | BI 1467335 3 mg Tablet (Japanese) | BI 1467335 6 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Caucasian)
Number analyzed (Participants) | 9 | 9 | 9 | 8
nanomole*hour/Liter (nmol*h/L) | 21.4 (51.1) | 117 (33.7) | 1120 (24.1) | 721 (86.2)
Statistical Analysis 1: Comparison: BI 1467335 3 mg Tablet (Japanese) vs BI 1467335 6 mg Tablet (Japanese) vs BI 1467335 10 mg Tablet (Japanese); This was non confirmatory testing on Day 28 (after multiple doses). Dose proportionality of tablets for AUC0-24,28 was analysed in Japanese subjects; Test type: Other; Slope = 3.2440, 95% CI 2-sided [2.8793 to 3.6087], Standard Error of Mean 0.1771 — [estimate comment as in outcome 2, analysis 1]; Standard error of mean is standard error of slope

5. Secondary Outcome: Cmax,28
Description: Maximum measured concentration of BI 1467335 in plasma following administration of 28th dose (Cmax,28).
Time Frame: as for outcome 4
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 3 mg Tablet (Japanese) | BI 1467335 6 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Caucasian)
Number analyzed (Participants) | 9 | 9 | 9 | 8
nanomole/Liter (nmol/L) | 13.2 (58.4) | 57.2 (35.1) | 159 (19.9) | 124 (41.8)
Statistical Analysis 1: Comparison: BI 1467335 3 mg Tablet (Japanese) vs BI 1467335 6 mg Tablet (Japanese) vs BI 1467335 10 mg Tablet (Japanese); This was non confirmatory testing on Day 28 (after multiple doses). Dose proportionality of tablets for Cmax,28 was analysed in Japanese subjects; Test type: Other; Slope = 2.0711, 95% CI 2-sided [1.7663 to 2.3760], Standard Error of Mean 0.1480 — [estimate comment as in outcome 2, analysis 1]; Standard error of mean is standard error of slope

ADVERSE EVENTS:
Time Frame: From first day of trial medication intake until end of trial, up to 48 days.
Description: Treated Set (TS): All subjects who received at least 1 dose of trial medication.
Arm/Group | Placebo (Japanese) | BI 1467335 3 mg Tablet (Japanese) | BI 1467335 6 mg Tablet (Japanese) | BI 1467335 10 mg Tablet (Japanese) | Placebo (Caucasian) | BI 1467335 10 mg Tablet (Caucasian)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 5/9 | 2/9 | 3/9 | 0/3 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Japanese) (N=9) | BI 1467335 3 mg Tablet (Japanese) (N=9) | BI 1467335 6 mg Tablet (Japanese) (N=9) | BI 1467335 10 mg Tablet (Japanese) (N=9) | Placebo (Caucasian) (N=3) | BI 1467335 10 mg Tablet (Caucasian) (N=9)
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT03159455/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT03159455/SAP_001.pdf